CLINICAL TRIAL: NCT05732636
Title: Urdu Translation And Cross-Cultural Validation of the Foot And Ankle Disability Index for the Patients With Chronic Ankle Instability
Brief Title: Urdu Translation And Cross-Cultural Validation of the Foot And Ankle Disability Index
Status: Completed | Type: Observational
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Other Study IDs: sairaakbar0444
Record Dates: First submitted 2023-01-27; First posted 2023-02-17 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Ankle Disorders Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validation study — The whole protocol is divided into two stages: Urdu Translation and validation. Following steps were involved.
  1. First version (Forward Translation): Forward translation from the English to Urdu by two bilingual translators (Version 1)
  2. Second Version: Three experts compared the original FADI with urdu version of FADI.
  3. Backward translation: Version 2 was translated Back in English by an independent translator.
  4. Third Version: was finalized after tracking differences in forward and backward translation.
  5. Final Version: of Urdu FADI was used on Chronic Ankle Instability patients.
  Foot and Ankle Disability Index(FADI) Urdu version was introduced and the patients were asked to fill FADI Urdu version. The questionnaire was filled again by the same participants after one week to assess the test retest reliability.

SUMMARY:
The goal of this Cross-cultural validation study is to Urdu translate and cross-cultural validation of Foot and Ankle Disability Index for the Patients with Chronic Ankle Instability. The main question it aims to answer was:

• To Translate Foot and Ankle Disability Index in Urdu and to find out the Validity and Reliability for Patients with Chronic Ankle Instability.

Data collection procedure would be, FADI Urdu version was introduced and the patients were asked to fill FADI Urdu version. The questionnaire was filled again by the same participants after one week to assess the test retest reliability. Questionnaire was conducted to have the best result. After the ethical approval, participants who meet the inclusion criteria and who were free from exclusion criteria were explained about the objectives of this study. Only those who gave consent were included in the study.

DETAILED DESCRIPTION:
The foot and ankle are common sources of pain and disability, with approximately 2 million people in the United States per year affected by foot pain. As many as 25% of sports injuries have been attributed to the foot or ankle, with ankle sprains accounting for up to 45% of all injuries in some sports. The Foot and Ankle Disability Index (FADI) were designed to assess functional limitations related to foot and ankle conditions. Therefore, it is used to assess the patients with chronic ankle instability. The FADI was originally developed in English. It has been translated and validated in Italian languages and showed excellent reliability and responsiveness. To cross culturally validate the FADI in Urdu, the FADI will be translated in Urdu to assess the chronic ankle instability patients to check the instability. Convenience sampling technique will be used in this study. A study will be conducted at Pakistan Sports Board Lahore including 10 athletes for 1st stage and 50 Athelets in 2nd stage. The aim of this study was to translate FADI in Urdu and to find out the validity and reliability of Urdu version of FADI in patients with chronic ankle instability. Reliability and validity of FADI in Urdu version was evaluated by calculating Cronbach's alpha, intra-class correlation co-efficient and Pearson/ spearman rank correlation co-efficient. SPSS 25 was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* A history of ankle sprain with pain and/or limping for more than 1 day,
* Chronic weakness, pain, or instability that they attributed to the initial injury
* Giving way in the last 6 months.
* Able to read Urdu Language

Exclusion Criteria:

* Bilateral ankle instability
* History of ankle fracture
* Ankle injury within 3 months of participation
* History of anterior cruciate ligament injury
* History of balance disorder
* Current participation in supervised physical rehabilitation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Athletes at Pakistan Sports Board with Chronic Ankle Instability.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Urdu version of Foot and Ankle Disability Index | at Day 7
  The Foot and Ankle Disability Index is a 34-item questionnaire divided into two subscales: the Foot and Ankle Disability Index and the Foot and Ankle Disability Index Sport. The FADI has 26 items, and the FADI Sport has 8. The FADI contains 4 pain related items and 22 activity related items. The FADI Sport contains 8 activity related items. It assesses more difficult tasks that are essential to sport. The FADI Sport is unique in that it is a population-specific subscale designed for athletes. It is designed to address this need by detecting deficits in higher functioning subjects.
Foot and ankle ability measure (FAAM) | at Day 7
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. It is a 29-item questionnaire divided into two subscales: the Foot and Ankle Ability Measure, 21-item Activities of Daily Living Subscale and the Foot and Ankle Ability Measure, 8-item Sports Subscale. Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. Item score totals, which range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale, were transformed to percentage scores. Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Akbar Bodla, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board Lahore, Lahore, Punjab Province, Pakistan